CLINICAL TRIAL: NCT00944398
Title: Evaluation of the Use of Plasma Zinc Concentration for Assessing the Impact of Targeted and Mass Zinc Fortification Programs
Brief Title: Impact of Targeted Zinc Fortification Programs on Plasma Zinc Concentration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Helen Keller International (Other); Cheikh Anta Diop University, Senegal (Other); Global Alliance for Improved Nutrition (Other)
Responsible Party: Prof. Kenneth H. Brown, Helen Keller International
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 200817275; 107008
Record Dates: First submitted 2009-07-21; First posted 2009-07-23 (Estimated); Last update posted 2010-02-19 (Estimated); Status verified 2010-02

CONDITIONS: Zinc Deficiency
Keywords: Zinc fortification; Plasma zinc concentration; Assessment of zinc status
MeSH Terms: interventions — Zinc Sulfate; Vitamin B Complex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Zinc fortified group (Experimental): Daily consumption of zinc-fortified complementary food
  Interventions: Dietary Supplement: Zinc fortified food; Other: Placebo supplement
- Non-fortified group (Placebo Comparator): Daily consumption of non-fortified complementary food and placebo supplement.
  Interventions: Other: Placebo supplement; Dietary Supplement: Non-fortified food
- Zinc supplement group (Experimental): Daily consumption of zinc supplement and non-fortified complementary food.
  Interventions: Dietary Supplement: Zinc supplement; Dietary Supplement: Non-fortified food

INTERVENTIONS:
Dietary Supplement: Zinc fortified food — Daily consumption
  Other Names: Provital, CoAID
  Arms: Zinc fortified group
Dietary Supplement: Zinc supplement — Liquid supplement containing zinc sulfate
  Other Names: Zinc sulfate and B vitamins, DSM
  Arms: Zinc supplement group
Other: Placebo supplement — Liquid placebo supplement
  Other Names: B vitamins, DSM
  Arms: Non-fortified group; Zinc fortified group
Dietary Supplement: Non-fortified food — Non-fortified complementary food.
  Other Names: Provital, CoAID
  Arms: Non-fortified group; Zinc supplement group

SUMMARY:
The purpose of the study is to evaluate the use of plasma zinc concentration for assessing the impact of targeted zinc fortification programs.

DETAILED DESCRIPTION:
The objectives of the present study are to determine whether plasma zinc concentration changes in response to additional zinc consumption, as provided by zinc-fortified cereal-based complementary foods fed to young children. The following specific steps will be completed:

1. Zinc-fortified complementary foods and breads prepared from zinc-fortified cereal flours will be developed with assistance from experts in food technology.
2. A two-week feeding trial will be implemented to assess the change in plasma zinc concentration among young children who receive: a) the zinc-fortified cereal porridge and a liquid vitamin preparation between meals; b) a non-zinc-fortified cereal porridge and a liquid vitamin preparation between meals [negative control group]; or c) a non-zinc-fortified cereal porridge and a zinc-containing liquid vitamin preparation between meals [positive control group].

ELIGIBILITY:
Inclusion Criteria:

* apparently healthy

Exclusion Criteria:

* severe malnutrition
* severe anemia

Ages: 12 Months to 17 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 98 (Actual)
Dates: Start 2009-01; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Plasma zinc concentration | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth H Brown, MD, Principal Investigator — University of California, Davis
Locations (1):
- Helen Keller International, Dakar, Senegal

REFERENCES:
- [Derived] Lo NB, Aaron GJ, Hess SY, Dossou NI, Guiro AT, Wade S, Brown KH. Plasma zinc concentration responds to short-term zinc supplementation, but not zinc fortification, in young children in Senegal1,2. Am J Clin Nutr. 2011 Jun;93(6):1348-55. doi: 10.3945/ajcn.111.012278. Epub 2011 Apr 13. PMID 21490143